CLINICAL TRIAL: NCT06749106
Title: Plaque Imaging in Routine Care to Detect Intraplaque Hemorrhage
Acronym: PARADE
Status: Recruiting | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: LMU Klinikum - Department of Neuroradiology (Unknown); LMU Klinikum - Department of Neurology (Unknown)
Responsible Party: Principal Investigator, Martin Dichgans, Prof. Dr. med. Martin Dichgans, Ludwig-Maximilians - University of Munich
Other Study IDs: PARADE
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Acute Ischemic Stroke
Keywords: plaque imaging; plaque vulnerability; cryptogenic stroke; routine care; stroke etiology; recurrent stroke; intraplaque hemorrhage; IPH; acute ischemic stroke; AIS
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- acute ischemic stroke: Patients with acute ischemic stroke, who received non-contrast carotid MRI for routine diagnostic work-up

SUMMARY:
The aim of this study is to investigate the association between intraplaque hemorrhage (IPH) detected by non-contrast magnetic resonance imaging (MRI) of the carotid artery in routine clinical practice and ipsilateral acute ischemic events. The investigators' overarching aim is to determine whether this sequence aids the diagnostic work-up of stroke patients.

For this purpose, the investigators set up a prospective single-center longitudinal observational study with one year follow-up. In addition, this study will analyze retrospectively obtained data collected through clinical routine.

DETAILED DESCRIPTION:
Stroke is one of the leading causes of death and the leading cause of permanent disability. Identifying the underlying etiology is crucial as secondary stroke prevention strategies vary depending on the cause of the stroke. However, in approximately 30% of patients, no clear etiology can be identified (cryptogenic stroke), preventing these patients from receiving targeted treatment.

Recent findings indicate that features of plaque vulnerability are associated with acute ischemic stroke which also applies to patients with cryptogenic stroke who have a carotid artery stenosis of less than 50%. Features of plaque vulnerability can be assessed by high-resolution carotid magnetic resonance imaging (MRI) which enables noninvasive detailed characterization of atherosclerotic carotid artery plaques. Hence, plaque imaging allows to detect vulnerable plaques and to further stratify stroke etiology. In addition, plaque imaging may identify patients with vulnerable plaques who are at risk for a recurrent ischemic stroke or TIA.

However, integrating multisequence high-resolution, contrast-enhanced MRI into the standard diagnostic workflow of acute stroke would prove difficult, thus calling for simpler imaging protocols. Unlike other features of plaque vulnerability, intraplaque hemorrhage (IPH) can be reliably detected by standard coils and conventional native black-blood fat-saturated T1-weighted sequences. Given the frequency of IPH, previous study results, and additional literature evidencing the importance of IPH as a marker for plaque vulnerability and risk of stroke recurrence, a single black-blood fat-saturated T1-weighted sequence was added to the MR imaging protocol for the diagnostic work-up of stroke patients at LMU hospital.

Patients with acute ischemic stroke, who received non-contrast carotid MRI for routine diagnostic work-up, will be asked whether they are willing to participate in a prospective, longitudinal study with telephone follow-up to assess recurrent ischemic stroke or TIA. In addition, this study will analyse retrospectively obtained data collected through clinical routine. These analyses will be done on all patients who received non-contrast carotid MRI for routine diagnostic work-up over the last years. This approach allows to estimate the prevalence of IPH in an unselected patient population.

In principle, the detection of IPH points towards the presence of an increased plaque vulnerability. However, it is unknown whether IPH can be reliably detected on routine clinical scans and whether information on the presence or absence of IPH should influence clinical decision making. Depending on the results, the outcome of this study might benefit future generations of patients by improving the diagnostic assignment to a specific stroke etiology and risk assessment with respect to recurrent vascular events.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute ischemic stroke
* Availability of non-contrast carotid MRI scans obtained through routine diagnostic work-up

Exclusion Criteria:

* Infarct in the posterior circulation or bilateral ischemic infarcts
* Time between symptom onset and non-contrast carotid MRI > 10 days
* Prior stenting of a carotid artery or carotid endarterectomy
* Age < 18 years
* Life expectancy < 1 year
* Inability to provide written informed consent

This eligibility criteria apply for the prospective part of the PARADE study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke, who received non-contrast carotid MRI for routine diagnostic work-up, will be asked whether they are willing to participate in a prospective, longitudinal study with telephone follow-up to assess recurrent ischemic stroke or TIA. Patients who are unable to provide informed consent for themselves, children and adolescents will not be recruited.
  Detailed eligibility criteria for the prospective longitudinal study are provided above.
  In addition, this study will analyse retrospectively obtained data collected through clinical routine: These analyses will be done on all patients who received non-contrast carotid MRI for routine diagnostic work-up over the last years. This approach allows to estimate the prevalence of IPH in an unselected patient population.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
intraplaque hemorrhage (IPH) | baseline
  presence of IPH as detected on routine non-contrast MRI

SECONDARY OUTCOMES:
recurrent ischemic stroke or TIA | 3 months, 12 months
  recurrent ischemic stroke or transient ischemic attack (TIA)
Plaque-RADS | baseline
  scoring plaque vulnerability according to the Plaque-RADS (Reporting and Data System) classification (score [1-4] with higher scores meaning higher plaque vulnerability) with all data available from clinical routine
Barthel Scale | baseline, 3 months, 12 months
  activities of daily living, assessed using the Barthel Scale (score [0-100] with lower scores meaning lower independence in activities of daily living)
modified Rankin Scale (mRS) | baseline, 3 months, 12 months
  modified Rankin Scale (mRS) as a functional global outcome scale measuring the level of disability after stroke (score [0-6] with higher scores meaning a worse outcome)
National Institutes of Health Stroke Scale (NIHSS) | baseline
  stroke severity, assessed using the National Institutes of Health Stroke Scale (NIHSS) (score [0-42] with higher scores meaning higher stroke severity)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Kopczak, MD, Principal Investigator — Institute for Stroke and Dementia Research
Locations (1):
- Institute for Stroke and Dementia Research, Munich, Germany

IPD SHARING:
Plan to Share IPD: Undecided
depending on the research proposal and the variables required